Red Blood Cell ATP Release and Vascular Function in Humans NCT03404843

May 19, 2018

## Fasudil Statistical Analysis Plan

All values are reported as mean ± SEM. All analyses were performed using R (R Core Team 2016, R Foundation for Statistical Computing, Vienna, Austria) with the Ime4, ImerTest, pbkrtest, and Ismeans packages. Age (young or older), drug (saline or fasudil), condition (rest or exercise intensity or hypoxia), and age×drug×condition for three-way repeated measures or age×drug for two-way repeated measures ANOVA were treated as fixed effects. In order to account for the crossover design, subject and subject×drug were in included in the model as random effects for the three-way repeated measures analyses and subject was included as a random effect for the two-way repeated measures analyses. When an interaction or main effect was found, appropriate pairwise comparisons were made and a Tukey test was included when necessary. Comparisons of variables relative to zero were tested using a one-tailed t-test, and differences in subject characteristics were tested using a two-tailed t-test. Comparisons between saline and fasudil were performed within age group and comparisons between young and old were performed within condition. Significance was set at P < 0.05.